CLINICAL TRIAL: NCT05822622
Title: Relationship Between Heart Failure With Preserved Ejection Fraction and Nonalcoholic Fatty Liver Disease.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Elsayed Khalifa, resident of internal medicine, Sohag University
Other Study IDs: Soh-Med-23-02-03
Record Dates: First submitted 2023-03-26; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Non Alcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF(heart failure with preserved ejection fraction): chronic heart failure with echocardiographic finding of LVEF (left ventricular ejection fraction) equal or more than 50% , diagnostic test :Abdominal ultrasound and transient elastography for detecting non alcoholic fatty liver disease .
  Interventions: Other: echocardiography
- NAFLD(non alcoholic fatty liver disease): ultrasound and transient elastographic finding of fatty liver disease, diagnostic test :echocardiography to determine heart failure with preserved ejection fraction .
  Interventions: Other: echocardiography

INTERVENTIONS:
Other: echocardiography — to determine finding of heart failure with preserved ejection fraction and non alcoholic fatty liver disease
  Other Names: abdominal ultrasound and transient elastography

SUMMARY:
The aim of our study to determine the demography, relation between patients with heart failure with preserved ejection fraction and those with nonalcoholic fatty liver disease in Sohag university hospital.

DETAILED DESCRIPTION:
type of the study cross sectional study to study the relationship between heart failure with preserved ejection fraction and nonalcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria: clinical diagnosis of heart failure with preserved ejection fraction.

clinical diagnosis of nonalcoholic fatty liver disease. -

Exclusion Criteria: rheumatic heart disease ,congenital heart disease , ischemic heart disease ,heart failure with reduced ejection fraction , hepatitis B virus , hepatitis C virus .

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients presented by heart failure with preserved ejection fraction and those with fatty liver disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-29 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
collection of results of echocardiography (those detect HFpEF) with abdominal ultrasound and transient elastography results (those detect NAFLD) and find relationship between the results. | up to 28 weeks.
  looking for relationship between echocardiographic findings (that detect heart failure with preserved ejection fraction) and finding in abdominal ultrasound and transient elastography (detection of nonalcoholic fatty liver disease) to detect the relationship between those two diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Aml K Ahmed, A professor, Study Chair — Sohag University; Alshimaa L Hamed, lecturer, Study Chair — Sohag University
Locations (2):
- Egypt (2):
  - Asmaa elsayed khalifa, Sohag, El Monshah
  - Asmaa E khalifa, Sohag

REFERENCES:
- [Result] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469